CLINICAL TRIAL: NCT05102968
Title: Using a Mobile APP to Support Home-based Rehabilitation for Patients With Rotator Cuff Tear After Arthroscopic Repair
Brief Title: The Effect of Self-rehabilitation Using Communication APP After Arthroscopic Surgery for Rotator Cuff Tear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Futing Huang, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS 18-CT12-15
Record Dates: First submitted 2021-10-01; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff tear; Arthroscopic surgery; Telerehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with mobile application (Active Comparator): Patients self-managed rehab exercise with a supportive mobile application
  Interventions: Behavioral: Home-based rehabilitation supporting with the mobile application
- Rehabilitation under supervision (Active Comparator): Patients received supervised physical therapy
  Interventions: Behavioral: Supervised rehabilitation by the therapist

INTERVENTIONS:
Behavioral: Home-based rehabilitation supporting with the mobile application — For patients with mobile application supportive rehabilitation, patients managed rehabilitation exercise by themselves after the surgery without supervision. Rehabilitation protocol and exercise instruction video were available in the application. Patient could communicate with the physician and therapist via the application.
  Other Names: Home exercise
  Arms: Rehabilitation with mobile application
Behavioral: Supervised rehabilitation by the therapist — For patients with therapist supervised rehabilitation, patients attended one-on-one instructions with a therapist (once a week at post-operative 2nd~12th week and once two weeks at post-operative 13th~24th week; totally 16 sessions in the 6-month rehabilitation program) and exercised under supervision at hospital. Subjects would receive additional sessions based on the rehabilitation progress. Subjects could cancel scheduled sessions by personal reasons. We provided telephone consultation without APP communication for subjects in the supervised group.
  Other Names: Supervised exercise
  Arms: Rehabilitation under supervision

SUMMARY:
The purpose of this study was to assess the clinical effect of a mobile application supporting home-based rehabilitation for the patients after arthroscopic rotator cuff repair. The investigators hypothesized the clinical results of the patients using a mobile application (APP) to support the home-based rehabilitation were comparable to the patients receiving the supervised rehabilitation.

This prospective randomized case-control study was approved by the institutional review board of the Kaohsiung Veteran General Hospital (IRB No. KSVGH18-CT12-15) prior to enroll any patients. Patients were recruited if they had a small to medium-sized full-thickness rotator cuff tear or, a Lafosse type II or III subscapularis tear diagnosed and then repaired under shoulder arthroscope. After the surgery, patients were randomized either to the home-based rehabilitation (the home group) or the hospital supervised rehabilitation (the supervised group).

In the home group, patients self-managed rehabilitation exercise without supervision. Rehabilitation were supportive with the APP. Patient could communicate with the physician via the APP. In the supervised group, patients attended one-on-one instructions with therapists and exercised under supervision at hospital.

Patients' characters were recorded. Peri-operative factors associated with rotator cuff healing were assessed. The active ROM (forward elevation, abduction, external and internal rotation), the visual analogue scale (VAS) pain scores, the American shoulder and elbow surgeon shoulder (ASES) scores and the modified Constant scores were recorded pre-operatively and post-operatively 3, 6, 12 and 24 months. The isometric shoulder strength was assessed with the hand-held dynamometer. The compliance of post-operative rehabilitation was evaluated not only from patients' self-reported logs but also by physicians at post-operatively 6, 12 and 24 weeks. Tendon integrity was evaluated with MRI scan at least 6 months after the index surgery. In the pilot study, we found a mean difference of 4 points and a standard deviation of 5.5 points in the modified Constant scores. Power analysis revealed a total sample size of 62 patients (31 patients in each group) would achieve a statistical power of 0.8 with a two-tailed level of 0.05 to detect significant differences. Statistical level of significance was defined as p<0.05.

DETAILED DESCRIPTION:
Introduction- Arthroscopic repair in the treatment of rotator cuff tear had been accepted wildly. It had been demonstrated that surgical management improved life quality and reduced economic burdens. However, joint stiffness and cuff re-tear, the two most common complications after arthroscopic cuff repair were concerned. Post-operative rehabilitation and its compliance are crucial for resilience. For rehabilitation, performing exercise too slowly caused joint stiffness, but too aggressively increased the risk of cuff re-tear. To prevent these complications, supervised physical therapy was advised after rotator cuff repair. However, the associated cost of rehabilitation under supervision exacerbated patients' financial burden. Home-based rehabilitation had been proposed and employed wildly, such as for the cardiopulmonary function after coronary artery disease, the ambulation training after joint replacement and the muscle strengthening after ACL reconstruction. In the conservative treatment of frozen shoulder and rotator cuff tear, patients with home-based physical therapy obtained comparable outcomes to supervised physical therapy. After arthroscopic rotator cuff repair, the clinical benefit of home-based rehabilitation was still controversial. In previous studies, supervised rehabilitation was not superior to home-based rehabilitation in long-term functional outcomes. However, some authors considered that the rehabilitation under supervision reduced the risk of cuff re-tear and joint stiffness. Furthermore, the patients who received the home-based rehabilitation supporting with a booklet or videotape had inferior compliance. For resolving the above-mentioned problems, supporting with a mobile application was possibly an alternative. It is a trend nowadays that telerehabilitation was assisted with mobile applications, such as for patients with stroke, spinal cord injury and musculoskeletal trauma. There was still lack of the literature about such rehabilitation method for the patients after arthroscopic rotator cuff repair. The purpose of this study was to assess the clinical effect of a mobile application supporting home-based rehabilitation for the patients after arthroscopic rotator cuff repair. The investigators hypothesized the clinical results of the patients using a mobile application to support the home-based rehabilitation were comparable to the patients receiving the supervised rehabilitation.

Patients Registries- This prospective randomized case-control study was approved by the institutional review board of the Kaohsiung Veteran General Hospital (IRB No. KSVGH18-CT12-15) prior to enroll any patients. Eligible patients were determined by the attending surgeon. After the surgery, a research assistant conducted the informed consent process before the enrollment in the study. Subjects were randomized either to the home-based rehabilitation (the home group) or the hospital supervised rehabilitation (the supervised group). Each patient was assigned a study number in a consecutive sequence. A randomization sequence using two variables was determined by the mobile application. The allocation of two rehabilitation modes according to the randomization sequence was designated to each subject in a sealed envelope. The therapist opened envelopes at the 1st day post-operatively.

Surgical procedures- Arthroscopic rotator cuff repair for all patients were performed by a single senior surgeon (F.H) at Kaohsiung Veteran General Hospital. Under general anesthesia, patients sit on the beach-chair. The posterior, posterolateral, lateral, and anterolateral portals were created. Intra-articular lesions including subscapularis and biceps long-head tendon were evaluated via the posterior viewing portal. For a Lafosse type II or III tear, subscapularis was repaired with one or two anchors under posterior visualization. Tenotomy, tenodesis or labrum repair for biceps lesions was performed according to labrum tear pattern, age, and functional demand. Rotator cuff lesion was addressed while viewing from the lateral portal. The dimension of involved cuff from anterior to posterior was measured with a probe. Single- or double-row repair was performed based on tear size and pattern. Acromioplasty or partial distal clavicle resection was performed if indicated.

Rehabilitation protocol- All patients received the one standard rehabilitation protocol and used the booklet that described the rehabilitation exercise in detail. The 6-month rehabilitation protocol consisted of four stages. The first stage was the immobilization phase that patients wear the arm sling for 2-4 weeks. The second stage was the ROM phase that patients started from passive to assisted-active ROM for 4-6 weeks. The third stage was the low-tensity training phase that patients allowed active ROM and isokinetic elastic-band exercise for 4-8 weeks. The fourth stage was the joint stabilization phase that patients focused on training the muscle for scapular stabilization and continued isokinetic exercise at least 2 months post-operatively. All patients were follow-up in the clinic every 4-6 weeks after the surgery. After the clinical visit, they were instructed by therapists to perform exercise at home while proceeding the next rehabilitation stage. The exercise program was adjusted according to the recovery status of each patient.

Intervention- In the home group, patients managed rehabilitation exercise by themselves after the surgery without supervision. Rehabilitation protocol and exercise instruction video were available in the APP. Patient could communicate with the physician and therapist via the APP. In the supervised group, subjects attended one-on-one instructions with a therapist (once a week at post-operative 2nd~12th week and once two weeks at post-operative 13th~24th week; totally 16 sessions in the 6-month rehabilitation program) and exercised under supervision at hospital. Subjects would receive additional sessions based on the rehabilitation progress. Subjects could cancel scheduled sessions by personal reasons. We provided telephone consultation without APP communication for subjects in the supervised group.

Outcome evaluation- Patients characters including age, sex, body mass index, arm dominance, trauma history, education background and functional demand were recorded. Peri-operative factors associated with rotator cuff healing were assessed. The active ROM (forward elevation, abduction, external and internal rotation), the visual analogue scale (VAS) pain scores, the American shoulder and elbow surgeon shoulder (ASES) scores and the modified Constant scores were recorded by a research assistant preoperatively and post-operatively 3, 6, 12 and 24 months. Biceps, subscapularis, infraspinatus, and supraspinatus index were measured post-operatively 3, 6, 12 and 24 months. The compliance of post-operative rehabilitation was assessed at post-operatively 6, 12 and 24 weeks. Tendon integrity was evaluated with MRI scan (a 1.5-T unit) at least 6 months after the surgery.

Sample size analysis and statistics methods- In the pilot study, the investigators found a mean difference of 4 points and a standard deviation of 5.5 points in the modified Constant scores. Power analysis revealed a total sample size of 62 patients (31 patients in each group) would achieve a statistical power of 0.8 with a two-tailed level of 0.05 to detect significant differences. All statistical analyses were performed using the SPSS (version 23; IBM, Armonk, NY). Categorical data between groups were compared with the Pearson's chi-squared test or Fisher's exact test. Comparisons of normally distributed continuous data with the independent t-test and non-normally distributed continuous data with the rank sum test were performed. The analysis of covariance was used to compare the subjective scores (the VAS pain scores, ASES scores and modified Constant scores) and objective outcomes (active ROM and muscle index) between two groups. Statistical level of significance was defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients had a small to medium-sized (less than 3 cm) full-thickness rotator cuff tear or, a Lafosse type II or III subscapularis tear diagnosed and repaired by shoulder arthroscope
* patients were willing to consent to post-operative rehabilitation randomization and commit to the two-year clinical follow-up period.

Exclusion Criteria:

* pre-operative shoulder stiffness (defined as passive forward elevation less than 100 degrees and external rotation loss over 50% comparing to the contralateral side)
* an intra-operative irreparable cuff tear
* a prior ipsilateral shoulder surgery
* a history of systemic auto-immune disease or septic arthritis of the ipsilateral shoulder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The modified Constant scores | post-op 6 months
  The Constant scores (the total score - 100 maximal points) included both physical examination findings of motion and strength (65 points) and patient-reported subjective evaluation of shoulder function (35 points) to analyze the function of normal and diseased shoulders. The scale consisted of several sections: pain (15 points), patient-reported function with activities of daily living (20 points), range of motion (40 points), and strength testing (25 points). Finally, the scores was normalized to the age and sex of the subject as the modified Constant scores. A higher score indicates better shoulder function.
The modified Constant scores | post-op 24 months
  The Constant scores (the total score - 100 maximal points) included both physical examination findings of motion and strength (65 points) and patient-reported subjective evaluation of shoulder function (35 points) to analyze the function of normal and diseased shoulders. The scale consisted of several sections: pain (15 points), patient-reported function with activities of daily living (20 points), range of motion (40 points), and strength testing (25 points). Finally, the scores was normalized to the age and sex of the subject as the modified Constant scores. A higher score indicates better shoulder function.

SECONDARY OUTCOMES:
The American shoulder and elbow surgeon shoulder (ASES) scores | post-op 6 months
  The ASES score contains a physician-rated and patient-rated section. The pain visual analog scale (VAS) and 10 functional questions are used to tabulate the reported ASES score. The total score - 100 maximum points - is weighted 50% for pain and 50% for function. The pain score (maximum 50 points) is calculated by subtracting the VAS from 10 and multiplying by five. The functional score is calculated from 10 questions(a scale from 0 to 3) for a maximal score of 50 points. The pain and functional portions are then summed to obtain the final ASES score. A higher score represent better function.
The American shoulder and elbow surgeon shoulder (ASES) scores | post-op 24 months
  The ASES score contains a physician-rated and patient-rated section. The pain visual analog scale (VAS) and 10 functional questions are used to tabulate the reported ASES score. The total score - 100 maximum points - is weighted 50% for pain and 50% for function. The pain score (maximum 50 points) is calculated by subtracting the VAS from 10 and multiplying by five. The functional score is calculated from 10 questions(a scale from 0 to 3) for a maximal score of 50 points. The pain and functional portions are then summed to obtain the final ASES score. A higher score represent better function.
The degree of active range of motion (ROM) of shoulder joint | post-op 6 months
  Regarding evaluation of the degree of active shoulder ROM, the angle for forward flexion, abduction, external rotation with the arm at the side was measured with a goniometer. Internal rotation was recorded by the maximal height achieved with the ipsilateral thumb when attempting to reach behind the back (ipsilateral thumb to the point of anatomic landmarks：0 points=lateral aspect of thigh, 2 points=behind buttock, 4 points=sacroiliac joint, 6 points=waist, 8 points=12th thoracic vertebrae, 10 points=inter-scapular level).
The degree of active range of motion (ROM) of shoulder joint | post-op 24 months
  Regarding evaluation of the degree of active shoulder ROM, the angle for forward flexion, abduction, external rotation with the arm at the side was measured with a goniometer. Internal rotation was recorded by the maximal height achieved with the ipsilateral thumb when attempting to reach behind the back (ipsilateral thumb to the point of anatomic landmarks：0 points=lateral aspect of thigh, 2 points=behind buttock, 4 points=sacroiliac joint, 6 points=waist, 8 points=12th thoracic vertebrae, 10 points=inter-scapular level).
The biceps, subscapularis, Infraspinatus and supraspinatus index | post-op 6 months
  Biceps, subscapularis, infraspinatus, and supraspinatus index were defined as the ratio of bilateral maximal isometric strength in a specific motion. The isometric strength was assessed with MicroFET hand-held dynamometer (MicroFET 2, Hogan Health Industries Inc., Biometrics, The Netherlands). Biceps strength was measured by the resistance of elbow flexion to 90 degrees with supinated forearm. Subscapularis strength was measured by the lift-off test in prone position. Infraspinatus and supraspinatus strength were measured by the resistance of shoulder external rotation and shoulder abduction respectively in lying side position. Subjects gradually increased the force and sustained in maximum for 3 seconds. For eliciting maximum strength, each muscle contraction was performed for 5 seconds and repeated two times with a 10-second interval.
The biceps, subscapularis, Infraspinatus and supraspinatus index | post-op 24 months
  Biceps, subscapularis, infraspinatus, and supraspinatus index were defined as the ratio of bilateral maximal isometric strength in a specific motion. The isometric strength was assessed with MicroFET hand-held dynamometer (MicroFET 2, Hogan Health Industries Inc., Biometrics, The Netherlands). Biceps strength was measured by the resistance of elbow flexion to 90 degrees with supinated forearm. Subscapularis strength was measured by the lift-off test in prone position. Infraspinatus and supraspinatus strength were measured by the resistance of shoulder external rotation and shoulder abduction respectively in lying side position. Subjects gradually increased the force and sustained in maximum for 3 seconds. For eliciting maximum strength, each muscle contraction was performed for 5 seconds and repeated two times with a 10-second interval.
The integrity of rotator cuff tendon | post-op 6 months
  Tendon integrity was evaluated with MRI scan (a 1.5-T unit) at least 6 months after the repair. The images were reviewed by the senior radiologist who was blinded to the rehabilitation group of patients. Tendon integrity was determined as "intact", "partial tear" and "complete tear", according to Sugaya's classification.

OTHER OUTCOMES:
The grade of compliance of post-operative rehabilitation | post-op 6 weeks
  The compliance of post-operative rehabilitation was evaluated not only from patients' self-reported logs but also by physicians at post-operatively 6 weeks. For patients, the log recorded the grade of home-exercise frequency as "high" (exercise 5-7 days per week), "intermediate" (exercise 2-4 days per week) and "low" (exercise 0-1 day per week). In the clinics, physicians questioned patients about the rehab-principle, activity, and frequency to assess of the compliance of doing home-exercise in three grades (high, intermediate, and low).
The grade of compliance of post-operative rehabilitation | post-op 12 weeks
  The compliance of post-operative rehabilitation was evaluated not only from patients' self-reported logs but also by physicians at post-operatively 12 weeks. For patients, the log recorded the grade of home-exercise frequency as "high" (exercise 5-7 days per week), "intermediate" (exercise 2-4 days per week) and "low" (exercise 0-1 day per week). In the clinics, physicians questioned patients about the rehab-principle, activity, and frequency to assess of the compliance of doing home-exercise in three grades (high, intermediate, and low).
The grade of compliance of post-operative rehabilitation | post-op 24 weeks
  The compliance of post-operative rehabilitation was evaluated not only from patients' self-reported logs but also by physicians at post-operatively 24 weeks. For patients, the log recorded the grade of home-exercise frequency as "high" (exercise 5-7 days per week), "intermediate" (exercise 2-4 days per week) and "low" (exercise 0-1 day per week). In the clinics, physicians questioned patients about the rehab-principle, activity, and frequency to assess of the compliance of doing home-exercise in three grades (high, intermediate, and low).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Lin, PhD, Study Director — Institute of Physical education, Health & Leisure Studies, National Cheng Kung University
Locations (1):
- Kaohsiung Veterns General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Background] Denard PJ, Ladermann A, Burkhart SS. Prevention and management of stiffness after arthroscopic rotator cuff repair: systematic review and implications for rotator cuff healing. Arthroscopy. 2011 Jun;27(6):842-8. doi: 10.1016/j.arthro.2011.01.013. PMID 21624680
- [Background] Thigpen CA, Shaffer MA, Gaunt BW, Leggin BG, Williams GR, Wilcox RB 3rd. The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Apr;25(4):521-35. doi: 10.1016/j.jse.2015.12.018. PMID 26995456
- [Background] Ross D, Maerz T, Lynch J, Norris S, Baker K, Anderson K. Rehabilitation following arthroscopic rotator cuff repair: a review of current literature. J Am Acad Orthop Surg. 2014 Jan;22(1):1-9. doi: 10.5435/JAAOS-22-01-1. PMID 24382874
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Ramey L, Osborne C, Kasitinon D, Juengst S. Apps and Mobile Health Technology in Rehabilitation: The Good, the Bad, and the Unknown. Phys Med Rehabil Clin N Am. 2019 May;30(2):485-497. doi: 10.1016/j.pmr.2018.12.001. Epub 2019 Mar 5. PMID 30954161
- [Background] Pires IM, Marques G, Garcia NM, Florez-Revuelta F, Ponciano V, Oniani S. A Research on the Classification and Applicability of the Mobile Health Applications. J Pers Med. 2020 Feb 27;10(1):11. doi: 10.3390/jpm10010011. PMID 32120849
- [Background] Alenabi T, Jackson M, Tetreault P, Begon M. Electromyographic activity in the immobilized shoulder musculature during ipsilateral elbow, wrist, and finger movements while wearing a shoulder orthosis. J Shoulder Elbow Surg. 2013 Oct;22(10):1400-7. doi: 10.1016/j.jse.2013.04.007. Epub 2013 Jun 14. PMID 23770113
- [Background] Cools AM, Dewitte V, Lanszweert F, Notebaert D, Roets A, Soetens B, Cagnie B, Witvrouw EE. Rehabilitation of scapular muscle balance: which exercises to prescribe? Am J Sports Med. 2007 Oct;35(10):1744-51. doi: 10.1177/0363546507303560. Epub 2007 Jul 2. PMID 17606671
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Katolik LI, Romeo AA, Cole BJ, Verma NN, Hayden JK, Bach BR. Normalization of the Constant score. J Shoulder Elbow Surg. 2005 May-Jun;14(3):279-85. doi: 10.1016/j.jse.2004.10.009. PMID 15889027
- [Background] Holmgren T, Oberg B, Sjoberg I, Johansson K. Supervised strengthening exercises versus home-based movement exercises after arthroscopic acromioplasty: a randomized clinical trial. J Rehabil Med. 2012 Jan;44(1):12-8. doi: 10.2340/16501977-0889. PMID 22124602
- [Result] Buker N, Akkaya S, Akkaya N, Gokalp O, Kavlak E, Ok N, Kiter AE, Kitis A. Comparison of effects of supervised physiotherapy and a standardized home program on functional status in patients with total knee arthroplasty: a prospective study. J Phys Ther Sci. 2014 Oct;26(10):1531-6. doi: 10.1589/jpts.26.1531. Epub 2014 Oct 28. PMID 25364104
- [Result] Grant JA, Mohtadi NG. Two- to 4-year follow-up to a comparison of home versus physical therapy-supervised rehabilitation programs after anterior cruciate ligament reconstruction. Am J Sports Med. 2010 Jul;38(7):1389-94. doi: 10.1177/0363546509359763. Epub 2010 Apr 1. PMID 20360607
- [Result] Krischak G, Gebhard F, Reichel H, Friemert B, Schneider F, Fisser C, Kaluscha R, Kraus M. A prospective randomized controlled trial comparing occupational therapy with home-based exercises in conservative treatment of rotator cuff tears. J Shoulder Elbow Surg. 2013 Sep;22(9):1173-9. doi: 10.1016/j.jse.2013.01.008. Epub 2013 Mar 22. PMID 23523073
- [Result] Roddey TS, Olson SL, Gartsman GM, Hanten WP, Cook KF. A randomized controlled trial comparing 2 instructional approaches to home exercise instruction following arthroscopic full-thickness rotator cuff repair surgery. J Orthop Sports Phys Ther. 2002 Nov;32(11):548-59. doi: 10.2519/jospt.2002.32.11.548. PMID 12449254
- [Result] Lisinski P, Huber J, Wilkosz P, Witkowska A, Wytrazek M, Samborski W, Zagloba A. Supervised versus uncontrolled rehabilitation of patients after rotator cuff repair-clinical and neurophysiological comparative study. Int J Artif Organs. 2012 Jan;35(1):45-54. doi: 10.5301/ijao.5000037. PMID 22287203
- [Result] Song SJ, Jeong TH, Moon JW, Park HV, Lee SY, Koh KH. Short-term Comparison of Supervised Rehabilitation and Home-based Rehabilitation for Earlier Recovery of Shoulder Motion, Pain, and Function after Rotator Cuff Repair. Clin Shoulder Elb. 2018 Mar 1;21(1):15-21. doi: 10.5397/cise.2018.21.1.15. eCollection 2018 Mar. PMID 33330146